CLINICAL TRIAL: NCT06665906
Title: Investigating the Use of A Patient Navigator to Address the Social Drivers of Health in the Management of Pain: A Pilot Study
Brief Title: Using a Patient Navigator to Address the Social Drivers of Health in the Management of Pain
Acronym: PANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00118893
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: daily pain; musculoskeletal pain; pain management
MeSH Terms: conditions — Pain; Musculoskeletal Pain; Agnosia | interventions — Social Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PainTrainer Followed by Social Intervention (Experimental): At study entry participants will receive web-based cognitive behavior therapy (PainTrainer) which is a self-guided program that contains 8 modules, lasting 30-40 minutes each and can be completed in 8 to 12 weeks. Each module teaches behavioral coping strategies for pain management and recommends practice exercises. At Week 12, social intervention will begin. Social intervention includes at least six phone call visits, plus or minus 4, with patient navigator to coordinate care.
  Interventions: Behavioral: Web-Based Cognitive Behavioral Therapy (PainTrainer); Behavioral: Social Intervention
- Social Intervention Followed by PainTrainer (Experimental): Participants will have social intervention at study entry. Social intervention includes at least six phone call visits, plus or minus 4, with patient navigator to coordinate care. At week 12, web-based cognitive behavior therapy (PainTrainer) will begin. PainTrainer is a self-guided program that contains 8 modules, lasting 30-40 minutes each and can be completed in 8 to 12 weeks. Each module teaches behavioral coping strategies for pain management and recommends practice exercises.
  Interventions: Behavioral: Web-Based Cognitive Behavioral Therapy (PainTrainer); Behavioral: Social Intervention
- PainTrainer Only (Experimental): At study entry participants will receive web-based cognitive behavior therapy (PainTrainer) which is a self-guided program that contains 8 modules, lasting 30-40 minutes each and can be completed in 8 to 12 weeks. Each module teaches behavioral coping strategies for pain management and recommends practice exercises.
  Interventions: Behavioral: Web-Based Cognitive Behavioral Therapy (PainTrainer)

INTERVENTIONS:
Behavioral: Web-Based Cognitive Behavioral Therapy (PainTrainer) — Self-guided program that contains 8 modules, lasting 30-40 minutes each and can be completed in 8 to 12 weeks. Each module teaches behavioral coping strategies for pain management and recommends practice exercises.
Behavioral: Social Intervention — At least six phone call visits, plus or minus 4, with patient navigator to coordinate care.
  Arms: PainTrainer Followed by Social Intervention; Social Intervention Followed by PainTrainer

SUMMARY:
The purpose of this study is to see if patients with chronic pain can improve how they manage their pain and daily function by working with a care manager and by learning pain coping skills from an online teaching tool.

DETAILED DESCRIPTION:
This study will determine the effects of patient navigator-delivered care coordination to address the major social drivers of health on pain-related outcomes. All participants will have access to web-based cognitive behavior therapy (PainTrainer) - a self-guided program that contains 8 modules, lasting 30-40 minutes each and can be completed in 8 to 12 weeks. Each module teaches behavioral coping strategies for pain management and recommends practice exercises. Some participants will also receive phone call visits with patient navigator to coordinate care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with daily pain for 3 months or longer
* Chronic daily musculoskeletal pain with Pain, Enjoyment, General Activity (PEG) Survey score >=4
* Primary care provider must be an Atrium provider
* Has at least one social driver of health: Financial insecurity, work and income, housing, food insecurity, safety, health literacy and at least one of the above, lack of social support and at least one of the above

Exclusion Criteria:

* Patients who have active cancer
* Cognitive impairment severe enough to preclude participation in a behavioral/lifestyle change program
* Live in a nursing home or inpatient treatment facility
* Unable to read and converse in English
* Those who are already connected to a patient navigator or nurse coordinator or social worker
* Planned elective surgery in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Rate of Participant Recruitment | Through study completion, on average 16 months
  Mean number of participants recruited each month. Formula for calculation is planned number of enrolled and randomized participants (30) divided by total number of months needed to recruit 30 participants. The higher the number, the faster the recruitment is (i.e., 30 participants divided by 15 months = 2 per month).
Rate of Participant Retention | Week 24
  Percentage of participants that completed study. Formula for calculation is number of participants that completed last study visit divided by the number of participants that were enrolled and randomized. Range 0 to 100%. The closer the percentage to 100%, the better is the follow-up rate (i.e., 26 completed week 24 study visit divided by 30 randomized participants = 86.6%).
Rate of Participant Engagement with Patient Navigator | Week 24
  Percentage of completed patient navigator phone calls. Formula for calculation is mean number of completed phone calls with the patient navigator divided by 6 scheduled phone calls. Range 0 to 100%. The higher the percentage, the better the rate of participant engagement with the patient navigator (i.e., 4 (average) number of completed phone calls divided by 6 scheduled calls = 66.6%).
Rate of Participant Engagement with PainTrainer | Week 24
  Percentage of completed PainTrainer modules. Formula for calculation is average number of completed PainTrainer modules divided by total number of modules (8). Range 0 to 100%. The closer the percentage to 100%, the better the rate of participant engagement with PainTrainer.

OTHER OUTCOMES:
Pain, Enjoyment, General Activity (PEG) Survey | Baseline, Week 12, Week 24
  Pain, Enjoyment, General Activity (PEG) Survey asks three questions about pain severity. Total score range is 0-30. Higher scores represent worse pain.
PROMIS Physical Functioning Short Form 6b | Baseline, Week 12, Week 24
  PROMIS Physical Functioning Short Form 6b is a 6 question survey about ability to perform basic physical daily activities. Total score range is 6-30. Higher score indicates better functioning.
PROMIS Sleep Disturbance 6a+ Sleep Duration | Baseline, Week 12, Week 24
  PROMIS Sleep Disturbance 6a+ Sleep Duration is a 13 question survey about sleep "over the past 7 days." Total score range from 13-65. Higher score indicates worse sleep and sleep related impairment.
Pain Catastrophizing Scale | Baseline, Week 12, Week 24
  Pain Catastrophizing Scale is a 6 question survey about how often a patient thinks catastrophically about their pain. Total scores range from 0-24. Higher score indicates increased thoughts and time spent on thinking about their pain.
PHQ-8 | Baseline, Week 12, Week 24
  PHQ-8 is an 8 question survey assessing depression severity. Total score range from 0-24. Higher score indicates more severe depression.
GAD-7 | Baseline, Week 12, Week 24
  GAD-7 is a 7 question survey assessing general anxiety "over the last 2 weeks." Total score range from 0-21. Higher score indicates more severe anxiety.
World Health Organization Quality of Life Survey | Baseline, Week 12, Week 24
  World Health Organization Quality of Life is a 2 question survey assessing patient perception of quality of life. Total score range from 2-10 for each question. Higher score indicates high quality of life perception.
UCLA Loneliness Scale | Baseline, Week 12, Week 24
  UCLA Loneliness Scale is a 3 question survey assessing social isolation. Total score range from 3-9. Higher score indicates higher level of social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ang, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT06665906/ICF_000.pdf